CLINICAL TRIAL: NCT01919905
Title: Fortification of Mozzarella Cheese With Vitamin D3: Effect of High Temperature Cooking and Bioavailability of Vitamin D3
Brief Title: Mozzarella Cheese Vitamin D and Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Toronto Metropolitan University (Other); George Brown College (Other)
Responsible Party: Principal Investigator, Reinhold Vieth, Clinical Biochemist, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: M2326
Record Dates: First submitted 2012-03-09; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Change in Serum 25 Hydroxyvitamin D Levels
Keywords: Mozzarella cheese fortification; Bioavailability of Vitamin D
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dose (Active Comparator): High dose vitamin D group receiving Mozzarella cheese/pizza with 28000 IU vitD/serving once a week
  Interventions: Dietary Supplement: Vitamin D
- Low dose (Placebo Comparator): Low dose vitamin D group receiving Mozzarella cheese/pizza with 200 IU vitD/serving once a week
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — High dose group receive 28000 IU vitamin D once a week Low dose group receive 200 IU vitamin D once a week

SUMMARY:
The purpose of this study is to evaluate the effect of heat on the bioavailability of vitamin D in industrially fortified mozzarella cheese baked with pizza.

DETAILED DESCRIPTION:
With a growing body of evidence, the Institute of Medicine (IOM) conducted a thorough review of all available evidence to publish a report on Dietary Reference Intakes (DRIs) for calcium and vitamin D. In the absence of adequate sun exposure, acquiring the new RDA of 600-800 IU/d for vitamin D through diet alone is difficult. There is a need to increase dietary sources of vitamin D for Canadians.

In a double blind, randomized trial, our objective was to assess the effect of high temperature pizza baking on the bioavailability of vitamin D3 fortified Mozzarella cheese. We tested the following hypotheses, set a priori: 1) vitamin D3 is bioavailable from pizza baked with fortified Mozzarella cheese and heat does not significantly break down vitamin D3; and 2) the change in serum 25(OH)D (from baseline to 10 wk) will be significantly greater in the high-dose vitamin D treated group (28000 IU/wk) compared to the low dose vitamin D-treated group (200 IU/wk).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females between ages 18-70 years

Exclusion Criteria:

* Use of vitamin D supplements in excess of 1000 IU/day
* A history of any medical disorder that might effect vitamin D or mineral metabolism
* Use of medications that could interfere with vitamin D metabolism
* Potential for sun exposure ( i.e travel to a sunny destination of use of tanning beds) within the month prior to or during the study
* History of hypercalcemia
* Unwillingness to return for follow up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Bioavailability of vitamin D fortified Mozzarella cheese after pizza baking | 2 months
  Blood 25(OH)D levels will be measured at baseline and at the end of the study between low dose vs. high dose vitamin D group.

SECONDARY OUTCOMES:
Monitoring dose safety | 2 months
  Monitor serum calcium, phosphate, creatinine, parathyroid hormone (PTH), as well as urine calcium, phosphate, and creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Vieth, Phd, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- George Brown College, Toronto, Ontario, Canada